CLINICAL TRIAL: NCT06071832
Title: Using Structured Video Chat to Improve Relationships Between Young Children and Remote Grandparents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lafayette College (Other)
Collaborators: University of South Dakota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: R15HD107457-01A1 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-10-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Family Members; Grandparents
Keywords: child development; cognitive development; grandparents; screen time; video chat; family relationships

STUDY DESIGN:
Intervention Model Description: In Aim 1, we will focus on the effects of structured video chat on child engagement and initiations of joint attention during video chat with grandparents.
  In Aim 2, we will determine whether structured video chat increases grandparents' enjoyment of the video chats and leads to greater feelings of closeness to their grandchild.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Structured Play Condition (Experimental): The following describes ONE intervention type with the following rationale. We chose to investigate shared book reading because it is a structured activity that is familiar, emotionally engaging, and supportive of general knowledge and language development. Adults report that shared reading is an important bonding activity that builds adult-child closeness through back- and-forth interactions. Importantly, the joint attention that occurs during shared book reading when adults and children share focus on the book may promote language and social emotional outcomes. Children are responsive and attentive during shared reading over video chat, but it is unknown whether a triadic interaction can be established during reading via video chat.
  Interventions: Other: Instructions for family Zoom session
- Structured Reading Condition (Experimental): The following describes ONE intervention type with the following rationale. For our structured play condition, we chose to investigate the activities of playing show and tell, imitating with objects, and drawing because these are common activities derived from lab-based video chat experiments with children, many of which are authored by the PI and Co-I.
  Interventions: Other: Instructions for family Zoom session
- Control Condition (Experimental): The control families will be asked to do video chat as usual, with no specific instructions.
  Interventions: Other: Instructions for family Zoom session

INTERVENTIONS:
Other: Instructions for family Zoom session — Within both play and reading conditions, we will manipulate the method of enacting the structured activities with the goal of facilitating different types of grandparent-initiated joint attention.

SUMMARY:
During the Coronavirus (COVID-19) pandemic many families are using video chat (e.g., Zoom) to maintain relationships with distant relatives, including grandparents. While 67% of all grandparents reported liking the idea of video chatting with their grandchildren, only 28% did so regularly. Increasing this percentage could significantly improve grandparent-grandchild relationships because the Preliminary Study 1 showed that video chat frequency is a strong predictor of grandparent's ratings of closeness to their grandchild, even after controlling for the geographic distance between them. The overall goal of the past, ongoing, and future research is to understand the cognitive and social developmental challenges of video chat in order to support its use with children. As the next step towards this goal, the investigators propose to directly compare two approaches to instructing grandparents on how to improve video chats between grandparents and young grandchildren (18-72 months of age). Families will use video chat without the involvement of researchers during each video chat. Parent-child- grandparent triads (n=180; the largest multi-session observational study of young children and video chat to date) will record 10 video chats under one of three randomly-assigned conditions: structured play, structured reading, or when given no instructions (control). The overall hypothesis is that structured video chat will increase children's engagement and joint attention (primary outcome measures), as well as grandparents' enjoyment of video chat and closeness with their grandchild (secondary outcome measures). The investigators will use detailed behavioral coding of the video recordings of these chats to objectively assess many of the outcome measures. The Preliminary Study 2 showed that structured video chat facilitates more positive social interactions. The proposed work extends the preliminary work because it translates laboratory methods to a complementary ecologically-valid approach in families' naturalistic environments. In Aim 1, the investigators will determine whether and for whom structured video chat improves child engagement and increases child-initiated screen- based joint attention during video chats between grandparents and grandchildren. In Aim 2, the investigators will determine whether structured video chat increases grandparents' enjoyment of the video chats and leads to greater feelings of closeness to their grandchild. Both principal investigators, who are at R15-eligible institutions, are well-qualified to complete the proposed work. Since 2017, they have published 9 papers on video chat, 12 papers on reading, and collaboratively completed 3 preliminary studies and 2 papers. They have mentored 77 undergraduate students, many of whom were co-authors on conference posters or presentations (37 students in total; 22 as a presenter) or journal articles. Importantly, 17 students came from underrepresented groups (BIPOC, first- generation in college, LGBT). A total of 47 are pursuing or have completed graduate work in health-related sciences, including 15 for doctoral degrees. The proposed work addresses a National Institute for Child Health & Development, Child Development and Behavior Branch's (CDBB) priority of advancing understanding of "Effects of Technology and Digital Media Use on Child and Adolescent Development."

DETAILED DESCRIPTION:
During the Coronavirus (COVID-19) pandemic, many families are using video chat (e.g., Zoom) to maintain relationships with distant relatives, including grandparents. Even before the pandemic, grandparent-grandchild relationships were challenging because >50% of grandparents had at least one grandchild who lived more than 200 miles away. While 67% of all grandparents reported liking the idea of video chatting with their grandchildren, only 28% did so regularly despite reporting technological self-efficacy and access to digital devices. Increasing this percentage could significantly improve grandparent-grandchild relationships because the Preliminary Study 1 showed that video chat frequency is a strong predictor of grandparent's ratings of closeness to their grandchild, even after controlling for the geographic distance between them. Video chat can be cognitively and socially challenging for young children. These challenges can lead to decreased child engagement during video chat, which in turn can decrease adult motivation to initiate video chat with (and therefore bond with) the child.

The overall goal of the investigators' past, ongoing, and future research is to understand the cognitive and social developmental challenges of video chat in order to support its use with children. As the next step towards this goal, the investigators propose to directly compare two approaches to instructing grandparents on how to improve video chats between grandparents and young grandchildren (18-72 months of age). Families will use video chat in a more naturalistic way than most prior research (i.e., without the involvement of researchers during each video chat). Parent-child-grandparent triads (n=180; the largest multi-session observational study of young children and video chat to date) will record 10 video chats under one of three randomly assigned conditions: structured play, structured reading, or when given no instructions (control). The overall hypothesis is that structured video chat will increase children's engagement and joint attention (primary outcome measures), as well as grandparents' enjoyment of video chat and closeness with their grandchild (secondary outcome measures). The investigators will use detailed behavioral coding of the video recordings of these chats to objectively assess many of the outcome measures. The Preliminary Study 2 showed that structured video chat facilitates more positive social interactions. The investigators will also examine the effects of three parallel methods of enacting the structured activities (grandparent-led, collaborative, and shared on-screen), which are designed to change the amount and type of joint attention that grandparents and grandchildren engage in during video chat. The Preliminary Study 3 indicates that during structured reading with a researcher over video chat, children engaged in more joint attention behaviors when they had their own copy of the book to follow along with versus when the book only appeared on the screen. The proposed work extends preliminary work because it translates previously-used laboratory methods to a complementary ecologically-valid approach.

Aim 1: Determine whether and for whom structured video chat improves child engagement and increases child-initiated screen-based joint attention during video chats between grandparents and grandchildren. Hypothesis 1.1: Both structured play and structured reading will increase engagement and joint attention compared to when no instructions are given. Hypothesis 1.2: The method of enacting activities within the structured reading and structured play conditions will promote different levels of engagement and different types of screen-based joint attention. Hypothesis 1.3: Child age will positively predict child engagement and joint attention across conditions. Hypothesis 1.4: The method of enacting activities will affect younger children's engagement and joint attention more than older children's. Exploratory Hypothesis 1.5: Structured play will increase engagement and joint attention more for younger children than older children, but older children will benefit more from structured reading. Hypothesis 1.6: Grandparent sensitivity will positively predict child engagement and joint attention, and this effect may be the strongest for younger children.

Aim 2: Determine whether structured video chat increases grandparents' enjoyment of the video chats and leads to greater feelings of closeness to their grandchild. Hypothesis 2.1: Grandparents will report an increase in enjoyment of video chats and greater feelings of closeness in the structured conditions compared to when no instructions are given. Hypothesis 2.2: The different methods of enacting activities within the structured conditions will promote different feelings of grandparent enjoyment and closeness. Hypothesis 2.3: Child age will predict grandparent closeness but not enjoyment.

Both principal investigators are at R15-eligible institutions, are well-qualified to oversee the proposed work. Since 2017, they have published 9 papers on video chat, 12 papers on shared reading, and collaboratively completed 3 preliminary studies and 2 papers. They have mentored 77 undergraduate students, many of whom were co-authors on conference posters or presentations (37 students total; 22 as a presenter) or journal articles (12 students). Importantly, 17 came from underrepresented groups (BIPOC, first-generation in college, LGBT). A total of 47 are pursuing or have completed graduate work in health-related sciences, including 18 for doctoral degrees. The proposed work will also address the National Institute for Child Health & Development, Child Development and Behavior Branch's (CDBB) priority of advancing understanding of "Effects of Technology and Digital Media Use on Child and Adolescent Development."

ELIGIBILITY:
Inclusion Criteria:

* have a child between the ages of 18 months and 5 years
* all parties speak English
* stable internet connection for all parties
* access to laptop, smart phone or tablet that can be used for Zoom interactions
* be able to hear to communicate effectively with partners in Zoom interactions
* see the screen well enough to communicate effectively on Zoom

Exclusion Criteria:

* does not meet any of the inclusion criteria

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Child engagement | Through study completion, an average of 2 months
  Frequency of the number of occurrences of smiles, nods, & on-topic verbalizations. To be measured by observing recordings of behavior.
Child initiation of within-screen joint attention | Through study completion, an average of 2 months
  Frequency of child's references to something in their own environment, paired with a look to the grandparent. e.g., child brings a toy to show grandparent. To be measured by observing recordings of behavior.
Child initiation of across-screen joint attention | Through study completion, an average of 2 months
  Frequency of child's direction of the grandparent's attention to an object or person on the other side of the screen, paired with a look to the grandparent. e.g., child points to her grandmother's dog. To be measured by observing recordings of behavior.
Grandparent Sensitivity | Through study completion, an average of 2 months
  Time-sampled in intervals of 30-seconds (coder gives a score for the sensitivity of each adult, based on that 30- second interval as one unit). Grandparent's accuracy in reading child signals, appropriate responsiveness to such signals, adult affect, awareness of timing, and flexibility to child's needs in the moment. Sensitivity will be coded following previously published criteria and will be a global rating that "emphasizes behavioral style rather than discrete behaviors" and accounts for the dyadic nature of sensitivity (child's needs affect parent's responses, and vice versa). To be measured by observing recordings of behavior.
Parental Involvement | Through study completion, an average of 2 months
  Frequency and duration of instances when the parent supports the child to engage with the grandparent, e.g., offers help. To be measured by observing recordings of behavior.

SECONDARY OUTCOMES:
Grandparent enjoyment | Through study completion, an average of 2 months
  Grandparents will be asked to self-report their enjoyment of the video chat on an Enjoyment scale, rated from 1 (not at all) to 5 (very much)
Grandparent closeness | Through study completion, an average of 2 months
  Grandparents will be asked to self-report their their closeness to the child on a Closeness scale, rated from 1 (strongly disagree) to 7 (strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren J Myers, Ph.D., Principal Investigator — Lafayette College
Locations (1):
- Lafayette College, Easton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data at the conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available in 2026 after our coding is complete.